CLINICAL TRIAL: NCT00804973
Title: A Safety, Tolerability, and Efficacy Study of LY2590443 in the Treatment of Acute Migraine Headache
Brief Title: Study in Participants With Acute Migraines Headaches
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to efficacy results of interim analysis
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 12258; I2W-MC-DMAB (Other: Eli Lilly)
Record Dates: First submitted 2008-12-05; First posted 2008-12-09 (Estimated); Results first posted 2020-05-19 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Migraine Headache
Keywords: Migraine; Headache
MeSH Terms: conditions — Migraine Disorders; Headache | interventions — Sumatriptan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: LY2590443; Drug: Placebo injection
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo injection; Drug: Placebo capsule
- 3 (Active Comparator)
  Interventions: Drug: Sumatriptan; Drug: Placebo capsule

INTERVENTIONS:
Drug: LY2590443 — 200 milligrams (mg) as four 50-mg capsules, oral, once
  Arms: 1
Drug: Placebo injection — saline solution, injection, once
  Arms: 1; 2
Drug: Sumatriptan — 6 milligrams (mg) injection (0.5 milliliter [mL] of 12 mg/mL solution), once
  Arms: 3
Drug: Placebo capsule — 4 capsules, once
  Arms: 2; 3

SUMMARY:
This is a Phase 2, multicenter, randomized, double-blind, placebo and active comparator-controlled study of LY2590443 in approximately 200 participants with migraines.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants between the ages of 18 and 65 years, inclusive.
* Participants who have migraine headaches, with or without aura (diagnosis according the International Classification of Headache Disorders-II), for at least 1 year.
* Participants who have had 2-8 migraine attacks on average per month for the last 3 months (but less than 15 headache days per month).
* Participants who are willing and able to comply with the study schedule and requirements.
* Participants who speak, read, and understand English sufficiently well and are willing to provide written informed consent.
* Participants who in the opinion of the principal investigator are in good general health.
* Venous access should be sufficient to allow blood sampling as per protocol.

Exclusion Criteria:

* Participants who do not or may not tolerate 5HT1 agonist treatments, with known hypersensitivity to sumatriptan (as discussed with the investigator).
* Female participants who have a positive pregnancy test at screening or pre- dose evaluation, or are breastfeeding.
* History or presence of significant medical illnesses as determined by the investigator.
* Participants with a current clinical diagnosis of major psychiatric disease.
* Regular use of known drugs of abuse; use of opiates for migraine rescue (no more than two times per month) is permissible.
* Blood donation of 500 milliliter (mL) or greater of whole blood products within 4 weeks of study commencement, during the study, or 4 weeks following the study.
* Investigator site personnel directly affiliated with this study and their immediate families. Immediate family is defined as a spouse, parent, child, or sibling, whether biological or legally adopted.
* Consumption of more than three units of alcohol per day where one unit is defined as a 12 ounces (oz) beer, 4 oz wine, or 2 oz of alcohol spirit liquor.
* Are unwilling or unable to comply with the use of a diary to directly record data from the participant.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2008-11; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (19):
- United States (19):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beverly Hills, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chula Vista, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fresno, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Garden Grove, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Imperial, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Diego, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Francisco, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santa Monica, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., West Palm Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chicago, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wellesley Hills, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ann Arbor, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mount Vernon, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., West Chester, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Philadelphia, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Memphis, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Austin, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Houston, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Norfolk, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- LY2590443: 200 milligrams (mg) administered once as four 50-mg capsules
- Sumatriptan: 6 milligrams (mg) administered once as an injection of 0.5 milliliter (mL) of 12 mg/mL solution
- Placebo: Administered once as 4 capsules or once as an injection of saline solution
Period: Overall Study
Arm/Group | LY2590443 | Sumatriptan | Placebo
Started | 40 | 40 | 40
Received at Least 1 Dose of Study Drug | 40 | 40 | 40
Completed | 40 | 40 | 40
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants who received at least 1 dose of study drug (LY2590443, sumatriptan, or placebo).
Groups:
- Total: Total of all reporting groups
Arm/Group | LY2590443 | Sumatriptan | Placebo | Total
Number analyzed (Participants) | 40 | 40 | 40 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.30 (12.40) | 39.53 (12.94) | 37.48 (10.58) | 39.10 (11.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 26 | 29 | 83
  Male | 12 | 14 | 11 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 7 | 15
  Not Hispanic or Latino | 36 | 36 | 33 | 105
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 3 | 3 | 1 | 7
  Black or African American | 10 | 10 | 7 | 27
  White | 25 | 24 | 29 | 78
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 1 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 40 | 40 | 40 | 120

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Headache Pain Free Response
Description: Participants were required to assess the presence of a headache and grade the intensity of the headache as "severe," "moderate," "mild," or "none." Headache pain free response was defined as the number of participants with a migraine pain intensity score of "none."
Time Frame: 2 hours after study drug administration
Population: All participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | LY2590443 | Sumatriptan | Placebo
Number analyzed (Participants) | 40 | 40 | 40
Participants | 6 | 12 | 6

2. Secondary Outcome: Number of Participants With Pain Free Response
Description: Participants were required to assess the presence of a headache and grade the intensity of the headache as "severe," "moderate", "mild," or "none." Pain free response was defined as the number of participants with a migraine pain intensity score of "none."
Time Frame: 30 minutes, 1 hour, 1.5 hours, 3 hours, and 4 hours after study drug administration
Population: All participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | LY2590443 | Sumatriptan | Placebo
Number analyzed (Participants) | 40 | 40 | 40
Participants
  30 Minutes Post-dose | 7 | 8 | 4
  1 Hour Post-dose | 1 | 5 | 2
  1.5 Hours Post-dose | 3 | 10 | 5
  3 Hours Post-dose | 14 | 19 | 13
  4 Hours Post-dose | 25 | 30 | 24

3. Secondary Outcome: Number of Participants With Pain Relief Response
Description: Participants were required to assess the presence of a headache and grade the intensity of the headache as "severe", "moderate," "mild," or "none." Pain relief response was defined as the number of participants with a migraine pain intensity score of "none."
Time Frame: 30 minutes, 1 hour, 1.5 hours, 2 hours, 3 hours, and 4 hours after study drug administration.
Population: All participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | LY2590443 | Sumatriptan | Placebo
Number analyzed (Participants) | 40 | 40 | 40
Participants
  30 Minutes Post-dose | 7 | 8 | 4
  1 Hour Post-dose | 11 | 14 | 12
  1.5 Hours Post-dose | 17 | 25 | 18
  2 Hours Post-dose | 22 | 31 | 24
  3 Hours Post-dose | 34 | 35 | 35
  4 Hours Post-dose | 38 | 39 | 34

4. Secondary Outcome: Number of Participants With Sustained Pain Relief Response
Description: Participants were required to assess the presence of a headache and grade the intensity of the headache as "severe," "moderate," "mild," or "none." Sustained pain relief response was defined as the number of participants with no return of a "moderate" or "severe" headache after pain went down to "mild" or "none" at 2 hours.
Time Frame: 24 and 48 hours after study drug administration
Population: All participants who received at least 1 dose of study drug and had Sustained Pain Relief Response data.
Measure: Count of Participants; unit: Participants
Arm/Group | LY2590443 | Sumatriptan | Placebo
Number analyzed (Participants) | 22 | 31 | 24
Participants
  Pain Relief at 24 Hrs Post-dose | 19 | 28 | 24
  Pain Relief at 48 Hrs Post-dose | 19 | 27 | 23

5. Secondary Outcome: Number of Participants With Recurrent Migraine Headache Within 24 or 48 Hours
Description: The time to headache recurrence is presented as the number of participants experiencing at least 1 recurring headache within 24 or 48 hours of receiving study drug.
Time Frame: Up to 24 and 48 hours after study drug administration
Population: All participants who received at least 1 dose of study drug with evaluable migraine recurrence data.
Measure: Count of Participants; unit: Participants
Arm/Group | LY2590443 | Sumatriptan | Placebo
Number analyzed (Participants) | 39 | 39 | 39
Participants
  24 Hours Post-dose: number analyzed (Participants) | 39 | 38 | 37
  24 Hours Post-dose | 2 | 2 | 4
  48 Hours Post-dose | 6 | 4 | 6

6. Secondary Outcome: Number of Participants With Nausea
Description: The number of participants reporting nausea as a migraine symptom
Time Frame: Pre-dose, 30 minutes, 1 hour, 1.5 hours, 2 hours, 3 hours, and 4 hours after study drug administration.
Population: All participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | LY2590443 | Sumatriptan | Placebo
Number analyzed (Participants) | 40 | 40 | 40
Participants
  Pre-Dose | 18 | 16 | 25
  30 Minutes Post-dose | 13 | 19 | 19
  1 Hour Post-dose | 13 | 13 | 12
  1.5 Hours Post-dose | 8 | 10 | 8
  2 Hours Post-dose | 8 | 8 | 6
  3 Hours Post-dose | 6 | 7 | 3
  4 Hours Post-dose | 4 | 4 | 2

7. Secondary Outcome: Number of Participants With Phonophobia
Description: The number of participants reporting phonophobia as a migraine symptom
Time Frame: Pre-dose, 30 minutes, 1 hour, 1.5 hours, 2 hours, 3 hours, and 4 hours after study drug administration.
Population: All participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | LY2590443 | Sumatriptan | Placebo
Number analyzed (Participants) | 40 | 40 | 40
Participants
  Pre-Dose | 28 | 33 | 31
  30 Minutes Post-dose | 24 | 25 | 26
  1 Hour Post-dose | 19 | 20 | 22
  1.5 Hours Post-dose | 15 | 18 | 16
  2 Hours Post-dose | 11 | 13 | 12
  3 Hours Post-dose | 6 | 3 | 5
  4 Hours Post-dose | 4 | 1 | 3

8. Secondary Outcome: Number of Participants With Photophobia
Description: The number of participants reporting photophobia as a migraine symptom
Time Frame: Pre-dose, 30 minutes, 1 hour, 1.5 hours, 2 hours, 3 hours, and 4 hours after study drug administration.
Population: All participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | LY2590443 | Sumatriptan | Placebo
Number analyzed (Participants) | 40 | 40 | 40
Participants
  Pre-Dose | 38 | 37 | 38
  30 Minutes Post-dose | 33 | 31 | 36
  1 Hour Post-dose | 31 | 28 | 31
  1.5 Hours Post-dose | 25 | 23 | 27
  2 Hours Post-dose | 22 | 19 | 24
  3 Hours Post-dose | 12 | 9 | 10
  4 Hours Post-dose | 6 | 4 | 6

9. Secondary Outcome: Number of Participants With Vomiting
Description: The number of participants reporting vomiting as a migraine symptom
Time Frame: Pre-dose, 30 minutes, 1 hour, 1.5 hours, 2 hours, 3 hours, and 4 hours after study drug administration.
Population: All participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | LY2590443 | Sumatriptan | Placebo
Number analyzed (Participants) | 40 | 40 | 40
Participants
  Pre-Dose | 1 | 1 | 2
  30 Minutes Post-dose | 0 | 2 | 1
  1 Hour Post-dose | 1 | 1 | 0
  1.5 Hours Post-dose | 1 | 1 | 0
  2 Hours Post-dose | 1 | 0 | 0
  3 Hours Post-dose | 0 | 0 | 0
  4 Hours Post-dose | 0 | 0 | 0

10. Secondary Outcome: Number of Participants With Sustained Pain Free Response
Description: Participants were required to assess the presence of a headache and grade the intensity of the headache as "severe," "moderate," "mild," or "none. Sustained pain free response was defined as the number of participants with no return of a "mild," "moderate" or "severe" headache after pain intensity went down to "none" at 2 hours.
Time Frame: 24 and 48 hours after study drug administration
Population: All participants who received at least 1 dose of study drug and had Sustained Pain Free Response data.
Measure: Count of Participants; unit: Participants
Arm/Group | LY2590443 | Sumatriptan | Placebo
Number analyzed (Participants) | 6 | 12 | 6
Participants
  Pain Free at 24 Hours Post-dose | 5 | 11 | 6
  Pain Free at 48 Hours Post-dose | 5 | 9 | 6

ADVERSE EVENTS:
Arm/Group | LY2590443 | Sumatriptan | Placebo
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 13/40 | 16/40 | 3/40
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2590443 (N=40) | Sumatriptan (N=40) | Placebo (N=40)
Somnolence (Nervous system disorders) | 6 (6) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 5 (5) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2) | 4 (4) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 4 (4) | 0 (0)
Burning sensation (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 2 (2) | 0 (0) — The Organ System includes "administration site conditions."

LIMITATIONS AND CAVEATS:
The study was terminated at the end of Part 1 (due to lack of efficacy). Part 2 was not enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days